CLINICAL TRIAL: NCT04971005
Title: A Randomised Controlled Trial to Compare Ocrelizumab or Alemtuzumab With Autologous Hematopoietic Stem Cell Transplantation (aHSCT) in High Inflammatory Multiple Sclerosis (COAST)
Brief Title: Ocrelizumab or Alemtuzumab Compared With Autologous Hematopoietic Stem Cell Transplantation in Multiple Sclerosis - a Phase-2 Randomised Controlled Trial
Acronym: COAST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment due to low acceptance of the control arm.
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Neovii Biotech (Industry); Clinical Trial Center North (CTC North GmbH & Co. KG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: inims-009
Record Dates: First submitted 2020-08-12; First posted 2021-07-21 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: autologous hematopoetic stem cell transplantation; alemtzumab; ocrelizumab; randomised controlled trial; aggressive highly active multiple sclerosis; no evidence of diseae activity (NEDA)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab; Alemtuzumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to control (ocrelizumab or alemtuzumab) or intervention (aHSCT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (aHSCT) (Experimental): Autologous Hematopoietic Stem Cell Transplantation. Mobilisation will be performed with 2 g/m2 cyclophosphamide and 10 μg/kg G-CSF from day 5 until apheresis is completed. Conditioning will be 200 mg/kg cyclo-phosphamide and Anti-T-lymphocyteglobuline (Grafalon®, Neovii) with cu-mulative doses of 20 mg/kg given on day +1 (10 mg/kg) and day +2 (10 mg/kg).
  Interventions: Drug: Autologous Hematopoietic Stem Cell Transplantation
- Control (Active Comparator): In the control arm patient and physician will decide which treatment to choose. Patients will be either treated with ocrelizumab according to the SmPC (600 mg every 6 months continuously) or with alemtuzumab according to the SmPC (12 mg/day for 5 consecutive days and again after 365 days for 3 days).
  Interventions: Drug: Ocrelizumab; Drug: Alemtuzumab

INTERVENTIONS:
Drug: Autologous Hematopoietic Stem Cell Transplantation — Autologous Hematopoietic Stem Cell Transplantation
  Arms: Intervention (aHSCT)
Drug: Ocrelizumab — 600 mg every 6 months continuously
  Arms: Control
Drug: Alemtuzumab — 12 mg/day for 5 consecutive days and again after 365 days for 3 days
  Arms: Control

SUMMARY:
A multicentre controlled phase II trial to compare the efficacy and safety of ocrelizumab or alemtuzumab and autologous Hematopoietic Stem Cell Transplantation (aHSCT). Active relapsing-remitting MS-Patients will be included and randomised to ocrelizumab or alemtuzumab versus aHSCT. Primary endpoint will be the time to treatment failure as assessed by failure of NEDA (no evidence of disease activity) as represented by: no expanded disability status scale (EDSS) progression, no relapse, no new T2 lesion and no Gd-enhancing lesion.

This trial offers the opportunity to gain further information about efficacy and safety of all treatments and will give new insights into the immunology of highly active RRMS.

DETAILED DESCRIPTION:
A rater-blinded multicentre randomised controlled phase II trial to compare the efficacy and safety of ocrelizumab or alemtuzumab and aHSCT. Active RRMS-Patients will be included and randomised to ocrelizumab or alemtuzumab versus aHSCT. Primary endpoint will be the time to treatment failure as assessed by failure of NEDA (no evidence of disease activity) as represented by: no expanded disability status scale (EDSS) progression, no relapse, no new T2 lesion and no Gd-enhancing lesion.

aHSCT appears highly efficacious in reducing inflammatory disease activity and relapses in active relapsing-remitting MS. Cohort data show a long-term stagnation of inflammatory disease activity for up to 10 years and more after aHSCT. However, efficacy data from randomised controlled trials comparing aHSCT with approved treatments are still lacking.

The best available data concerning disease activity in MS patients with a documented treatment failure are from the CARE-MS II trial. The rate of patients without clinical or radiological disease activity after 2 years was 32% with alemtuzumab. aHSCT trial data on absence of disease activity show NEDA rates between 70 and 90% after 2 years. Here we assume 40% and 80% after 2 years for the ocrelizumab/alemtuzumab and aHSCT groups, respectively.

For all three treatments, a potential long-term benefit has to be balanced with potentially harmful treatment related risks. A randomised controlled trial offers the opportunity to gain further information about efficacy and safety of all treatments and will give new insights into the immunology of high active RRMS.

ELIGIBILITY:
Inclusion Criteria (Based on CARE-MS-II3, guidelines and Rio-criteria for treatment failure):

* Written informed consent and agreement to comply to study protocol
* Age: 18-55 years
* EDSS: 0.0 - 6.0
* RRMS according to McDonald 2010
* < 10 years of disease course after symptom onset
* Active disease with one of the following treatment failures occur-ring not earlier than 6 months after initiation of an approved DMT
* 2 or more relapses within the last 12 months

or

* 1 relapse within the last 12 months and a Gd-enhancing lesion on MRI > 3 mm > 3 months before or after relapse onset or 2 new T2-lesions

or

* On-going signs of MRI activity in the last 6 months (either Gd-en-hancing of ≥ 3 mm lesion at any exam in the last year; or more than 5 new T2 lesions (≥ 3 mm)

or

* Patients stable under natalizumab but who have to stop treatment due to an increasing PML risk are defined as active, if a MRI within 6 months after termination of natalizumab shows new T2 or Gd-enhancing lesions and at least one other treatment fail-ure prior to natalizumab is documented.

Exclusion Criteria:

* Secondary or primary progressive MS
* Pregnancy, or other medical condition incompatible with aHSCT
* Any treatment or medical condition that, according to the haematologist / transplant specialist precludes the use of aHSCT
* John Cunningham virus (JCV) antibody index of > 1.5 in previ-ously natalizumab-treated patients, if a negative CSF JCV-PCR prior to screening is not available
* Relapse during 30 days before initiation of treatment. If a relapse occurs during this period and eligibility criteria are otherwise ful-filled, start of treatment will be delayed until at least 30 days after receiving steroids.
* Concurrent clinically significant (as determined by the investiga-tors and haematologist / transplant specialist) cardiac, immuno-logical, pulmonary, neurological, renal or other major disease such as:

  * Prominent cardial disease (Left ventricular ejection frac-tion (LVEF) < 40%, myocardial infarction or ischemia, un-controlled arrhythmias, pericardial effusion > 1 cm)
  * Cerebrovascular disease
  * Renal disease (creatinine clearance < 30 ml/min/m2)
  * Respiratory disease (DLCO < 40% predicted)
  * Active bleeding or clotting disease
  * History of human immunodeficiency virus (HIV) or posi-tive HIV antibody testing
  * Any uncontrolled acute or chronic infection, including HIV, hepatitis B surface antigen positivity and hepatitis C PCR positivity
  * Cancer except in situ cervix or cutaneous
* Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, men-tal, or social) that is likely to affect the patient returning for follow-up visits on schedule. Unwillingness to use contraception.
* Previous participation in this study, previous treatment with aHSCT or already both comparators
* Ongoing immunotherapy. Treatment with interferon or glati-rameracetate will need no wash-out. Treatment pause before oc-relizumab/alemtuzumab or aHSCT will be:

  * for dimethylfumarate and fingolimod: 8 weeks
  * for natalizumab: 8 weeks
  * for ocrelizumab: 12 weeks
  * for alemtuzumab: 12 months
  * for teriflunomide: 4 weeks after elimination with cholesty-ramine
  * for cladribine: 24 weeks
* Patients with cognitive impairments who are unable to provide written, informed consent prior to any testing under this protocol, including screening and baseline investigations that are not con-sidered part of routine patient care.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure as assessed by failure of NEDA (no evidence of disease activity) | through study completion, on average at least 2 years
  Time to treatment failure as assessed by failure of NEDA (no evidence of disease activity) during follow-up as defined by:
  * 3 months confirmed EDSS (Expanded disability status scale) progression
  * confirmed relapse
  * new/enlarging T2-hyperintense lesion on MRI (Magnetic resonance imaging)
  * any Gd-enhancing lesion on MRI

SECONDARY OUTCOMES:
Efficacy of treatment defined by EDSS | through study completion, on average at least 2 years
  EDSS change and EDSS improvement will be considered. EDSS improvement defined as confirmed improvement after 3 months
Efficacy of treatment defined by the annualized relapse rate | through study completion, on average at least 2 years
  calculated as number of relapses per year
Efficacy of treatment defined by the number of new T2 lesions | through study completion, on average at least 2 years
  calculated as cumulative number of new T2 lesions
Efficacy of treatment defined by the number of Gd-enhancing lesions | through study completion, on average at least 2 years
  calculated as cumulative number of GD-enhancing lesions
Efficacy of treatment defined by multiple sclerosis functional composite (MSFC) change | through study completion, on average at least 2 years
  based on summed up Z-scores for individual measures (SDMT, 9 HPT, 25 FWT)
Efficacy of treatment defined by Hamburg quality of life scale in MS (HAQUAMS) | through study completion, on average at least 2 years
  based on HAQUAMS sum score ratings (values between 1 and 5)
Efficacy of treatment defined by the Percentage Brain Volume Change (PBVC) | through study completion, on average at least 2 years
  Brain tissue volume (grey matter, white matter) will be evaluated on T1 weighted images to compute absolute percentage brain volume change
Efficacy of treatment defined by grey and white matter atrophy | through study completion, on average at least 2 years
  based on grey and white matter volume change evaluated on T1 weighted images
Rate of AE / SAE including NCI grade 3 and 4 non-haematological toxicities | through study completion, on average at least 2 years
  Safety of treatment defined by the rate of AE / SAE including NCI grade 3 and 4 non-haematological toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kröger, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department of Stem Cell Transplantation
Locations (2):
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Mannheim, Mannheim